CLINICAL TRIAL: NCT00175435
Title: Optimizing Hepatitis B Vaccine Response Through the Use of a Topical Immune Modulator
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of British Columbia (Other)
Responsible Party: Dr. Jan Dutz, University of British Columbia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: C05-0027
Record Dates: First submitted 2005-09-11; First posted 2005-09-15 (Estimated); Last update posted 2010-11-02 (Estimated); Status verified 2010-10

CONDITIONS: Hepatitis B
Keywords: Topical Immune Modulator; resiquimod gel; Hepatitis B booster response; Vaccine Evaluation; Prevention of Hepatitis B disease
MeSH Terms: conditions — Hepatitis B

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Experimental): 2 doses of HPV vaccine 0.5 mL. given IM with Topical Immune Modulator in 9-13 year-olds.
  Interventions: Biological: Resiquimod gel
- 2 (Active Comparator): 3 doses of HPV vaccine 0.5 mL given IM with Topical Immune Modulator in 9-13 year-olds.
  Interventions: Biological: Resiquimod gel
- 3 (Active Comparator): 3 doses HPV vaccine 0.5 mL given IM with Topical Immune Modulator in 16-26 year-olds.
  Interventions: Biological: Resiquimod gel

INTERVENTIONS:
Biological: Resiquimod gel — 3 doses HPV vaccine 0.5 mL given IM with Topical Immune Modulator
  Other Names: HPV vaccine - Gardasil
  Arms: 1
Biological: Resiquimod gel — 3 doses HPV vaccine 0.5 mL given IM with Topical Immune Modulator.
  Other Names: HPV vaccine = Gardasil
  Arms: 2
Biological: Resiquimod gel — 3 doses HPV vaccine 0.5 mL given IM with Topical Immune Modulator.
  Other Names: HPV vaccine = Gardasil
  Arms: 3

SUMMARY:
This study will look at what happens to the level of protection against hepatitis B (HB) disease if a 'helper' gel is applied to the skin over the injection site of a small dose of hepatitis B vaccine.

ELIGIBILITY:
Inclusion Criteria:

* Previously vaccinated with conventional hepatitis B vaccine series 10 or more years ago
* Generally healthy
* Is and has been free of HB disease and/or is negative to core antibody
* Known to have sero-converted to positive after vaccine series (without extra doses)
* Speaks and understands English adequately
* Available for all 4 visits within the designated timelines (30 days)
* No allergies to HB vaccine or components
* No blood or blood components within previous 6 months
* Not pregnant or breastfeeding

Ages: 19 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 39 (Actual)
Dates: Start 2005-08; Primary Completion 2007-04 (Actual); Study Completion 2007-04 (Actual)

PRIMARY OUTCOMES:
A single application of an immune modulating gel will enhance the protective response against hepatitis B disease when vaccination is given at the same time as gel as evidenced by increased HB antibody and T-cell response. | at 30 days after vaccination

SECONDARY OUTCOMES:
Minimal adverse effects to gel application as noted by laboratory assessment of liver enzyme and complete blood count (CBC) and physical assessment of the site/surrounding area and solicited local and general post vaccine events. | at 7 and 30 days post vaccine

CONTACTS AND LOCATIONS:
Overall Officials: Jan Dutz, MD, Principal Investigator — University of British Columbia
Locations (1):
- Vancouver General Hospital Vaccine Education Centre, Vancouver, British Columbia, Canada